CLINICAL TRIAL: NCT00895817
Title: Comparison of Aerosolized Swallowed Fluticasone to Esomeprazole for the Treatment of Eosinophilic Esophagitis
Brief Title: Fluticasone Versus Esomeprazole to Treat Eosinophilic Esophagitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Fouad J. Moawad, Principal Investigator, Walter Reed Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-14045
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Results first posted 2013-03-12 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Eosinophilic Esophagitis
Keywords: Eosinophilic esophagitis; acid reflux
MeSH Terms: conditions — Eosinophilic Esophagitis; Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Swallowed fluticasone (Active Comparator)
  Interventions: Drug: Swallowed fluticasone
- Esomeprazole (Active Comparator)
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Swallowed fluticasone — 440 µg twice daily for 8 weeks
  Arms: Swallowed fluticasone
Drug: Esomeprazole — 40 mg once daily for 8 weeks
  Arms: Esomeprazole

SUMMARY:
The purpose of this study is to assess the clinical efficacy of proton pump inhibitors in comparison to aerosolized swallowed steroids for the treatment of eosinophilic esophagitis (EE). EE is an increasingly recognized disorder that has been associated with dysphagia and food impaction. The presence of anatomical abnormalities in the esophagus such as longitudinal furrows, corrugated rings and a narrow caliber esophagus with friable mucosa are classic endoscopic findings. Diagnosis is established with the histologic finding of large numbers (> 15) of eosinophils per high power field. The underlying pathologic mechanism remains poorly understood but food allergies and aeroallergens have been implicated. It is well known that gastroesophageal reflux disease (GERD) may cause esophageal eosinophilia, but it is unclear whether a complex relationship exists between GERD and EE, as recent data suggests. Furthermore, a large number of patients with clinical presentations and endoscopic findings highly suggestive of EE which is confirmed on histology are responding favorably to proton pump inhibitors.

The aims of the study are to (1) compare the clinical efficacy of aerosolized swallowed Fluticasone to Esomeprazole for the treatment of eosinophilic esophagitis, (2) determine whether proton pump inhibitors are effective in the treatment of eosinophilic esophagitis, (3) determine the number of patients with eosinophilic esophagitis that have coexisting gastroesophageal reflux disease, and (4) correlate change in eosinophil count to improvement in symptoms before and after therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established diagnosis of EE defined as > 20 eosinophils/HPF in the setting of dysphagia or food impaction.
* Males and females age > 18 years of age.
* Ability to undergo ambulatory pH monitoring.
* DEERS (Defense Enrollment Eligibility Reporting System) eligible.
* Willingness to take a one month holiday from a PPI or steroids if they have been prescribed this prior to enrollment.
* Willingness to participate and have additional biopsies taken during endoscopy and answer a questionnaire.

Exclusion Criteria:

* Patients < 18 years of age.
* Inability to give consent.
* Inability to undergo endoscopy or contraindications to endoscopy. Any medical condition or disorder (including drug allergies), which would preclude the use of conscious sedation or the ability to tolerate upper endoscopy.
* Contraindications to proton pump inhibitors or steroids.
* Inability to accurately fill out a short questionnaire.
* Pregnant females. A urine beta human chorionic gonadotropin (BHCG) prior to endoscopy will be offered to all female patients of child bearing potential (exceptions include post-menopausal, hysterectomy or bilateral tubal ligation). Positive BHCG results will prevent enrollment.
* Known coagulation abnormalities, thrombocytopenia and patients on coumadin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fouad J Moawad, M.D., Principal Investigator — Walter Reed Army Medical Center
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with symptoms of esophageal dysfunction were recruited from the GI clinic of Walter Reed Army Medical Center. Recruitment dates were from 2008-2010.
Pre-assignment Details: Subjects with a confirmed diagnosis of EE based on symptoms and tissue biopsies were offered enrollment.All subject underwent 24-hour pH studies to stratify GERD positive and GERD negative. A computer generated list of random numbers was then used to separate patients into two equal treatment groups (esomeprazole and fluticasone proprionate).
Groups:
- Esomeprazole: Esomeprazole : 40 mg once daily for 8 weeks
- Swallowed Fluticasone: Swallowed fluticasone : 440 µg twice daily for 8 weeks
Period: Overall Study
Arm/Group | Esomeprazole | Swallowed Fluticasone
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole | Swallowed Fluticasone | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38 (10) | 38 (10) | 38 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 19 | 19 | 38
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Responded
Description: Histologic resolution of esophageal eosinophilia. Response is defined as achieving < 7 eosinophils/high power field in both the proximal and distal esophagus.
Time Frame: 8 weeks
Population: Sample size estimation was based on the assumptions:10% of the EE patients will respond to PPI compared to 55% of patients treated with steroids. Controlling the probability of a Type I error at alpha=0.05, a sample of 38 patients in the treatment groups (19 in each arm) will have 80% power to detect a difference in treatment response of 45%.
Measure: Number; unit: participants
Arm/Group | Esomeprazole | Swallowed Fluticasone
Number analyzed (Participants) | 21 | 21
participants | 7 | 4

2. Secondary Outcome: Symptom Score
Description: Using a validated questionnaire, symptoms will be assessed at baseline and following therapy.
Time Frame: 8 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Endoscopic Change
Description: Following therapy, resolution of EE findings will be assessed.
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Esomeprazole | Swallowed Fluticasone
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No